CLINICAL TRIAL: NCT00112281
Title: A Phase III International, Multi-Center, Prospective, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Nitric Oxide Synthase Inhibition With Tilarginine Acetate Injection in Patients With Cardiogenic Shock Complicating Acute Myocardial Infarction, or the TRIUMPH Trial
Brief Title: A Study of the Safety and Efficacy of Nitric Oxide Reduction in Patients With Cardiogenic Shock After a Heart Attack
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Arginox Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARG-CS3-001
Record Dates: First submitted 2005-06-01; First posted 2005-06-02 (Estimated); Last update posted 2006-08-04 (Estimated); Status verified 2005-05

CONDITIONS: Shock, Cardiogenic
Keywords: shock, cardiogenic, "myocardial infarction"
MeSH Terms: conditions — Shock, Cardiogenic; Shock; Myocardial Infarction

INTERVENTIONS:
Drug: Tilarginine Acetate Injection intravenous infusion

SUMMARY:
Tilarginine Acetate Injection is a new type of drug that temporarily stops the body from making a bodily substance called nitric oxide. The body may produce excess nitric oxide following severe heart damage leading to shock. During a heart attack, and especially after a blocked artery causing the heart attack is reopened, a large amount of nitric oxide is released into the heart muscle and into the blood. Normally small amounts of nitric oxide are good for the heart and blood vessels. However, when released in large amounts, such as during a heart attack, it may be harmful, by adding to the damage of the heart attack and lowering the heart's ability to pump blood to the body. It may cause blood pressure to be lowered and reduce the amount of blood flow to the body's vital organs. This may interfere with the body's organs being able to do their work. If Tilarginine Acetate Injection can stop extra nitric oxide from being made, the performance of the heart and blood flow to the organs may get better, which may result in the improvement of symptoms. The purpose of this study (TRIUMPH) is to investigate the safety and effectiveness of Tilarginine Acetate Injection compared to placebo (an inactive fluid that has no effect on the body but looks exactly like the medication being studied). The study will help determine whether Tilarginine Acetate Injection, by temporarily lowering the amount of nitric oxide released into the vital organs can improve blood pressure and the blood flow to the body's organs.

DETAILED DESCRIPTION:
An estimated 120,000 to 160,000 patients annually are diagnosed with cardiogenic shock (CS) in North America and Europe. CS complicates approximately 5-14% of all cases of acute myocardial infarction (AMI) and is the most common cause of death in patients hospitalized with AMI. Cardiogenic shock developing during the course of AMI is the end result of a pathophysiological cycle secondary to a sudden and significant decrease in cardiac contractility due to infarction, ischemia, and stunning of large myocardial segments. It is not anticipated that further advances in reperfusion or revascularization therapy will have a significant additional impact on survival in patients with CS. Modalities that protect the myocardium during ischemia and reperfusion are likely to be the next major advance in improving outcome in the setting of acute myocardial infarction (MI), especially in patients with large infarcts complicated by shock. Preliminary studies investigating nitric oxide synthase (NOS) inhibition suggest that improvements in cardiovascular function and survival are possible by limiting formation of toxic NO. The primary objective of the TRIUMPH study is to establish the efficacy of Tilarginine Acetate Injection compared to placebo in reducing all cause mortality at 30 days post randomization in patients with cardiogenic shock complicating acute myocardial infarction (MI). Safety objectives of this study include an evaluation of adverse events and serious adverse events, and key laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed myocardial infarction (heart attack)
* Confirmed persistent cardiogenic shock
* Confirmed patency of the infarct related artery (heart attack artery has been opened through the use of a blood clot dissolving drug or a balloon or angioplasty heart procedure)
* Less than 24 hour duration of cardiogenic shock (the time since the heart attack occurred and the artery was opened must be less than 24 hours)

Exclusion Criteria:

* Infection
* Other cause of shock (not heart attack)
* Shock due to heart valve disease
* Severe heart valve disease
* Right sided heart failure
* Shock due to arrhythmia (irregular heart rhythm)
* Severe kidney disease
* Aortic dissection (tear in aorta)
* Adult respiratory distress syndrome (ARDS) (severe lung inflammation)
* Severe brain damage
* Severe irreversible multi-system failure (failure of multiple body organs)
* Major chest or abdominal surgical procedure within 30 days except if prior CABG and reocclusion occurs
* Primary pulmonary hypertension (high blood pressure in the arteries of the lungs)
* Age younger than 18 years
* Requirement for emergency coronary artery bypass grafting (CABG) or infarct-related artery occlusion (heart attack artery completely blocked)
* Ongoing or recent participation in another clinical trial of an investigational drug
* Prior enrollment in this study or rapid resolution of cardiogenic shock before treatment (shock gets better before study starts)
* Positive pregnancy test in women who are of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658
Dates: Start 2005-05; Study Completion 2007-01

PRIMARY OUTCOMES:
All cause mortality at 30 days post randomization

SECONDARY OUTCOMES:
Number of patients demonstrating resolution of cardiogenic shock compared to placebo
The duration of cardiogenic shock compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Judith S. Hochman, M.D., Study Chair — NYU Langone Health
Locations (102):
- United States (83):
  - The Heart Group, PC, Mobile, Alabama
  - Sparks Regional Medical Center, Fort Smith, Arizona
  - Banner Baywood Heart Hospital, Mesa, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Central Arkansas Cardiovascular Research Group (CACRG), Little Rock, Arkansas
  - Los Angeles Cardiology Associates, Los Angeles, California
  - University of Southern California, LAC + USC Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Desert Cardiology, Rancho Mirage, California
  - Mercy General Hospital, Sacramento, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Christiana Care Health Services, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Cardiovascular Research Center, Atlantis, Florida
  - Watson Clinic, LLP, Lakeland, Florida
  - Health First Clinical Research Institute, Melbourne, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Mt. Sinai Medical Center, Miami, Florida
  - Mediquest Research Group, Ocala, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Heart Care Midwest, Peoria, Illinois
  - Trinity Medical Center, Rock Island, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Iowa Health, Des Moines, Des Moines, Iowa
  - Iowa Heart Centre, Des Moines, Iowa
  - University of Iowa Hospital, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Northeast Cardiology Associates, Bangor, Maine
  - Maine Medical Center, Portland, Maine
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Interventional Cardiovascular Research - Lahey Clinic, Burlington, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Fallon Cardiology - St. Vincent Hospital, Worchester, Massachusetts
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Nisus Research at Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's Duluth Clinic Health System, Duluth, Minnesota
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - BryanLGH Heart Institute, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper Health System, Camden, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Lenox Hill Heart and Vascular Institute of New York, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Rochester Cardio-Pulmonary Group, P.C., Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Cardiology Associates of Schenectady, Schenectady, New York
  - Mission Hospitals, Asheville, North Carolina
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Sanger Clinic, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - LeBauer Cardiovascular Research, Greensboro, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MidWest Cardiology Research Foundation, Columbus, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Providence Heart & Vascular Institute, Portland, Oregon
  - The Heart Care Group, Allentown, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Guthrie Clinic, Sayre, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - South Carolina Heart Center, Columbia, South Carolina
  - Johnson City Medical Center, Johnson City, Tennessee
  - St. Thomas Cardiology Consultants, Nashville, Tennessee
  - Ben Taub General Hospital, Baylor College of Medicine, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Texas Medical School, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Fletcher Allen Healthcare, Burlington, Vermont
- Canada (19):
  - Calgary Heart Centre Alberta, Calgary, Alberta
  - Royal Alexandria Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver Hospital and Health Sciences Centre, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - NB Heart Centre, Saint John, New Brunswick
  - Cardiology Research - QEII Health Science Centre, Halifax, Nova Scotia
  - QEII Health Science Centre - Cardiology Research, Halifax, Nova Scotia
  - Hamilton Health Sciences, General Site, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Trilium Health Centre, Mississauga, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa, Ottawa, Ontario
  - St. Michael's Hospital Toronto, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Quebec Heart Institute, Québec, Quebec

REFERENCES:
- [Derived] TRIUMPH Investigators; Alexander JH, Reynolds HR, Stebbins AL, Dzavik V, Harrington RA, Van de Werf F, Hochman JS. Effect of tilarginine acetate in patients with acute myocardial infarction and cardiogenic shock: the TRIUMPH randomized controlled trial. JAMA. 2007 Apr 18;297(15):1657-66. doi: 10.1001/jama.297.15.joc70035. Epub 2007 Mar 26. PMID 17387132